CLINICAL TRIAL: NCT06382987
Title: Registry of Psoriasis Health Outcomes: A Longitudinal Real-world Collaboration (RePhlect) - A Real-World, Prospective, Observational Study of the Comparative Effectiveness of Deucravacitinib in Adults With Plaque Psoriasis in Japan
Brief Title: A Study of the Comparative Effectiveness of Deucravacitinib in Adults With Plaque Psoriasis in Japan (RePhlect)
Acronym: RePhlect
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1124
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — deucravacitinib; apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants that have initiated deucravacitinib treatment
  Interventions: Drug: Deucravacitinib
- Participants that have initiated apremilast treatment
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Deucravacitinib — According to the product label
  Groups: Participants that have initiated deucravacitinib treatment
Drug: Apremilast — According to the product label
  Groups: Participants that have initiated apremilast treatment

SUMMARY:
This is a prospective, observational, real-world study of adult participants in Japan with physician-reported diagnosis of plaque psoriasis treated with deucravacitinib or apremilast.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adult participants aged 18 years old or older
* Physician-reported diagnosis of plaque psoriasis
* Newly initiating deucravacitinib or apremilast according to the label
* Participants who have signed informed consent

Exclusion Criteria:

* Participants currently participating in or planning to participate in an interventional clinical trial
* Patients enrolled in deucravacitinib post-marketing surveillance study (ClinicalTrial.gov ID: NCT05633264)
* Previous treatment experience with the treatment of interest (e.g. patients who have history of apremilast will not be eligible to be enrolled in apremilast arm of the study and similar for deucravacitinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include Japanese adults with a physician-reported diagnosis of plaque psoriasis who start treated with either deucravacitinib or apremilast. Study participants will be enrolled from Japanese Dermatological Association (JDA)-certified hospitals and clinics that are allowed to prescribe molecular targeted agents for patients with psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in percent Body Surface Area (BSA) involved affected by plaque psoriasis from baseline to follow up in participants treated with deucravacitinib. | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieved Physician's Global Assessment (PGA) of 0/1 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieved Absolute Psoriasis Area and Severity Index (aPASI) of ≤2 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieved Dermatology Life Quality Index (DLQI) of 0 /1 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Participant duration of treatment (time difference between date of treatment initiation to date of discontinuation) | 1 month, 3 months, 6 months and every 6 months up to 5 years

SECONDARY OUTCOMES:
Change in percent Body Surface Area (BSA) involved affected by plaque psoriasis from baseline to follow up in participants treated with deucravacitinib or apremilast | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieved Dermatology Life Quality Index (DLQI) of 0/1 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Participant duration of treatment (time difference between date of treatment initiation to date of discontinuation) from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants treated with deucravacitinib with a change in Physician's Global Assessment (PGA) from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants treated with deucravacitinib with a change in Dermatology Life Quality Index (DLQI) from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants achieving a Dermatology Life Quality Index (DLQI) score of ≤5 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve a Psoriasis Area Severity Index (PASI) response of 75 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve a Psoriasis Area Severity Index (PASI) response of 90 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve an absolute Psoriasis Area Severity Index (aPASI) score ≤5 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve an absolute Psoriasis Area Severity Index (aPASI) score ≤3 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve a National Psoriasis Foundation (NPF) Acceptable Body Surface Area response from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve an absolute scalp-specific Physician's Global Assessment (ss-PGA) of 0/1 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve an absolute Physician's Global Assessment-Fingernail (PGA-F) of 0/1 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years
Number of participants who achieve an absolute Palmoplantar Physician's Global Assessment (pp-PGA) of 0/1 from baseline to follow-up | 1 month, 3 months, 6 months and every 6 months up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Mebix. Inc., Minato-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts